CLINICAL TRIAL: NCT02136550
Title: Smoking Cessation on the Human Airway: Mucus Secretion, Inflammatory and Proteomic Profile in Nasal Lavage and miRNAs in Blood
Brief Title: Smoking Cessation on the Human Airway: Mucus Secretion, Inflammatory and Proteomic Profile in Nose and miRNAs in Blood
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Naomi Kondo Nakagawa, Associate Professor of Physiotherapy, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CEP 147/13; FAPESP 2013/13598-1 (Other Grant/Funding Number: FAPESP 2013/13598-1)
Record Dates: First submitted 2014-05-06; First posted 2014-05-13 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Smoking; Smoking Cessation
Keywords: smoking; smoking cessation; mucociliary clearance; proteomics; miRNA
MeSH Terms: conditions — Smoking; Smoking Cessation

STUDY DESIGN:
Intervention Model Description: Subjects that entered in the Smoking Cessation Program at Institute Dante Pazzanese of Cardiology State of Sao Paulo
Masking Description: Fluid analysis and other physical measurements
Oversight: Data Monitoring Committee: No

ARMS (1):
- Smoking cessation (Experimental): 36 smokers will participate in the study and will be evaluated at baseline, 6 months e 12 months of the smoking cessation program. If they quit the program, they will be asked to continue the study.
  Interventions: Behavioral: Smoking cessation

INTERVENTIONS:
Behavioral: Smoking cessation — Smoking cessation is a program that gives all the support to the subject: orientation, medications, exams, etc

SUMMARY:
Smoking cessation improves health conditions with reduction of the risk factors for cardiovascular and respiratory disease, as functional capacity and quality of life. Smoking cessation has positive effects on the miRNAs regulation, however, genomics has been little explored. Smoking and aging induces changes miRNAs. Among the changes in airway epithelial cells, miR-125 called attention because it is enrolled in the suppression of ERBB7 (tirosin kinase receptors), a codified sequence of the growth factor receptor (EGFR) frequently expressed in cancer. The reduction of miR-125 expression may reduce cancer suppression resulting in cancer development. Other miRNA changes can be observed, such as miR-218 that were found in smokers airway epithelial cells as in MiR-15b that were found in lung tissue of COPD smokers. These miRNAs participated in the signalling pathway of TGF-β enrolled in leukocyte migration and cell proliferation. The investigators hypothesize that smoking cessation has a role in the regulation or reduction in the genetic changes smoking-induced. The investigators will assess the subject genomic profile at the baseline, 6 months and 12 months after smoking cessation.

DETAILED DESCRIPTION:
After agreement with the written informed consent, 36 volunteers, male and female, aged between 18 and 70 years will be recruited at Medical School University of Sao Paulo and in the Ambulatory of Smoking Cessation Program of the Clinics Hospital. Exclusion criteria are inability to taste saccharin, nasal surgery, respiratory infection in the previous 30 days to the enrollement into the study. All volunteers will be assessed at Basal, 6 months and 12 months. The present study aims to assess the effects of smoking cessation on the airway defense mechanism, airway inflammation and genomics (miRNAs) in humans by using (a) saccharin transit time test to assess mucociliary clearance; (b) mucus physical properties; (c) EBC pH; (d) Nasal lavage pH, cellularity,cytokines (IL-1β, TGF-β, TNF-α, IL-4, IL-6, IL-8, IL-10, IL-13, MPO, MUC5AC, cotinine, proteomics, (e) lung function; (f) genomics (miRNAs) and (g) quality of life with rhinosinusitis questionnaire (SNOT20), sleep disturbances questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* 36 subjects, male or female, aged between 18 and 70 years recruited at Medical School University of Sao Paulo and the Smoking Cessation Program of the Clinics Hospital

Exclusion Criteria:

* inability to taste saccharin, nasal surgery, infection in the last 30 days (before the study)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-12 (Actual); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
miRNAs expression | PParticipants will be followed for the duration of the cessation program, an expected average of 6 months
  Blood sample will be collected in paxgene tube (BD do Brasil, SP, Brasil). MicroRNAs will be extracted from the blood samples by using PAXgene blood miRNA kit (Qiagen Inc., Valencia, USA). PCR Array will be customized (Custom miScript miRNA PCR Array, Qiagen Inc., Valencia, USA) for the miRNAs analysis. The fluorescence signal will be detected by RotorGene (Qiagen Inc., Valencia, USA).

SECONDARY OUTCOMES:
saccharin transit time test | Participants will be followed for the duration of the cessation program, an expected average of 6 months
  We evaluate the nasal MCC by measuring nasal saccharine transport time (STT). The subject is asked to avoid alcohol, tea and coffee for 6 hours and to eat or drink nothing for 2 hours before the measurements. The STT assessment is performed in a quiet room at a temperature of 21-22ºC and relative humidity of 63-71%. Subjects sat in a chair and are asked to maintain regular breathing, to avoid deep breathing, coughing, sneezing, sniffing or talking during STT measurements. Twenty-five µg saccharin particles are deposited 2 cm from the anterior end of the non-obstructed nostril and the timer is stopped at the first perception of sweet taste. The maximum delay between the deposition and perception is set at 60 minutes for non-detection.
Airway acidification by exhaled breath condensate pH | Participants will be followed for the duration of the cessation program, an expected average of 6 months
  The EBC is obtained as previously described. At the start of EBC collection, all subjects rinse their mouths with distilled water and are instructed to swallow saliva as necessary and to hold a slight head extension (approximately 15o). The EBC sample is collected over 15 min of quiet and normal breathings (regular tidal volumes and respiratory rate) through a mouthpiece that is connected to a collector device with dry ice (-20 °C). The total EBC (2.0-2.5 ml) is immediately divided and transferred to sterile 500 μl polypropylene tubes. One aliquot is immediately used for pH measurements. The remaining EBC sample aliquots are coded (for blinding purposes) and stored for a maximum of 4 weeks at -80°C for the determination of cytokine levels.
Quality of life by St George Questionnaire | Participants will be followed for the duration of the cessation program, an expected average of 6 months
  This is a questionnaire validate for Brazilian population to assess the quality of life of individuals with chronic respiratory problems (de Souza et al, 2000)
inflammation in the upper airway by analysis of nasal lavage | Participants will be followed for the duration of the cessation program, an expected average of 6 months
  Celularity and determination of TNF-α, IL-1beta, IL1-RA, IL-4, IL-5, IL-6, IL-8, IL-9, IL-10, IL-13, IL-17, MPO, G-CSF, MUC5AC and cotinine (multiplex bead assay and ELISA) in nasal lavage. Celularity: the cell pellet is resuspended in one milliliter of phosphate buffer saline solution (PBS). Thereafter, 20 µl of the mixed solution is added to a Neubauer chamber, and the cells are counted using a 400x light microscope (Olympus CH2, Olympus America Inc., Palo Alto, USA). For differential cell counts, 100 µl of the mixed solution is centrifuged (96 g, 25°C, 6 min) to obtain a slide with two areas of cells that are stained with hematoxylin and eosin. Differential cell counts are performed with the aid of a 1000x light microscope (Olympus CH2, Olympus America Inc., Palo Alto, USA) by two different observers.
Upper airways symptoms by SNOT20 questionnaire | Participants will be followed for the duration of the cessation program, an expected average of 6 months
  This is a questionnaire that aims to assess quality of life of patients with chronic upper airways symptoms
sleep quality by Pittsburg questionnaire | Participants will be followed for the duration of the cessation program, an expected average of 6 months
  It is a questionnaire to assess the quality of sleep (basically 6 questions)

CONTACTS AND LOCATIONS:
Overall Officials: Paulo HN Saldiva, Professor, Study Director — University of Sao Paulo Medical School; Naomi K. Nakagawa, Professor, Principal Investigator — University of Sao Paulo Medical School
Locations (1):
- Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Utiyama DM, Yoshida CT, Goto DM, de Santana Carvalho T, de Paula Santos U, Koczulla AR, Saldiva PH, Nakagawa NK. The effects of smoking and smoking cessation on nasal mucociliary clearance, mucus properties and inflammation. Clinics (Sao Paulo). 2016 Jul;71(6):344-50. doi: 10.6061/clinics/2016(06)10. PMID 27438569